CLINICAL TRIAL: NCT02421835
Title: Olive Leaf Extract as Part of a Healthy Lifestyle in the Reduction of Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Olive Leaf Extract as Part of a Healthy Lifestyle in the Reduction of Blood Pressure, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLE Chronic Study 2015
Record Dates: First submitted 2015-04-10; First posted 2015-04-21 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Pre Hypertension
MeSH Terms: conditions — Prehypertension | interventions — olive leaf extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo control (Placebo Comparator): 2 capsules of 350 mg maltodextrin to be consumed daily for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Olive leaf extract (Active Comparator): 2 capsules of 350 mg olive leaf extract equivalent 132 mg of oleuropein in olive leaf extract to be consumed daily for 12 weeks
  Interventions: Dietary Supplement: Olive leaf extract
- Physical activity (Placebo Comparator): 2 capsules of 350 mg maltodextrin to be consumed daily combined with gradually increase physical activity levels over 12 weeks
  Interventions: Dietary Supplement: Placebo
- Physical activity and olive leaf extract (Active Comparator): 2 capsules of 350 mg olive leaf extract equivalent 132 mg of oleuropein in olive leaf extract to be consumed daily combined with gradually increase physical activity levels over 12 weeks
  Interventions: Dietary Supplement: Olive leaf extract

INTERVENTIONS:
Dietary Supplement: Olive leaf extract — 132 mg of oleuropein per day suspended in olive leaf extract 700 mg
  Arms: Olive leaf extract; Physical activity and olive leaf extract
Dietary Supplement: Placebo — 700 mg Maltodextrin per day
  Other Names: Maltodextrin
  Arms: Physical activity; Placebo control

SUMMARY:
Hypertension affects about 30% of the United Kingdom population and is causally implicated in the aetiology of renal disease, cardiovascular disease and stroke. Ageing, obesity, a poor diet and low levels of physical activity are all risk factors. Studies have shown that adherence to a Mediterranean diet is protective against hypertension and its associated morbidities; olive oil is believed to be a key beneficially bioactive component of that diet. As a source of lipids olive oil is an unremarkable blend of monounsaturated, polyunsaturated and saturated fatty acids; it is however rich in phenolic compounds, principally oleuropein and hydroxytyrosol, which may be of benefit to health. A recent randomised intervention trial in predominantly hypertensive volunteers showed that adherence to a Mediterranean diet supplemented with extra virgin olive oil, reduced blood pressure and other measures of cardiovascular disease risk. Olive phenolics can be extracted cheaply from the waste products of olive oil manufacture, such as the plant leaf and these are used as dietary supplements. In intervention studies in hypertensive or borderline hypertensive patients, olive leaf extract consumption has been shown to reduce blood pressure.

Another intervention with established efficacy for improving blood pressure is to increase physical activity. The 'Start Active, Stay Active', Chief Medical Officers report on physical activity recommends that adults achieve 150 minutes of moderate intensity physical activity per week, while data in that report suggest that fewer than 40% of adult men and 30% of adult women achieve these targets. Adherence to the physical activity guidelines may in fact be much worse in sub-sections of the population at higher risk of hypertension.

From a public health perspective, holistic guidelines for the prevention of hypertension, or its early diagnosis and management, based around a healthy diet and lifestyle are preferable to pharmaceutical intervention. Lifestyle interventions are economically favourable and they come with fewer side effects and perhaps wider health benefits than antihypertensive drugs.

The aim of the study is to evidence the synergistic benefits of consuming plant (and specifically olive) phenolics alongside achieving the recommended guidelines for physical activity in individuals with elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* 25-70y
* BMI >25kg/m2
* Not having suffered a myocardial infarction/stroke in the past 12 months
* Not diabetic (diagnosed or fasting glucose > 7 mmol/l) or suffer from other endocrine disorders
* Not suffering from renal or bowel disease or have a history of cholestatic liver or pancreatitis
* Not on drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* No history of alcohol misuse
* Not planning or on a weight reducing regime
* Not taking any fish oil, fatty acid or vitamin and mineral supplements
* Non smokers

Exclusion Criteria:

* Use of antibiotics within the previous 6 months
* History of alcohol or drug abuse
* Intake of any experimental drug within 4 weeks of the start of the study
* Excessive alcohol consumption (more than 21 units/wk male, 15 units/wk female)
* Females who are breast-feeding, may be pregnant, or of child-bearing potential and not using effective contraceptive precautions
* Have had recently (in the last 5 years) major surgery, which might limit participation in, or completion of, the study.
* On drug treatment for high blood fats, high blood pressure and blood clotting.
* Physical or mental diseases that are likely to limit participation or completion of the study

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure measured via 24 hour ambulatory blood pressure monitors | 12 weeks
  measured using the ScanMed Oscillometric Ambulatory blood pressure deviceVolunteers will be asked to wear the device which will be programmed to record BP measurements every 30 minutes during the day (7am-10pm) and every hour by night (10pm-7am)

SECONDARY OUTCOMES:
Average plasma glucose concentration | 12 weeks
  a measure of chronic blood sugar control) by measuring of glycated haemoglobin (HbA1c)
Vascular function assessed by pulse wave velocity (PWV) | 12 weeks
Plasma biomarkers of endothelial function including nitric oxide, vascular cell adhesion molecule (VCAM), Inter-Cellular Adhesion Molecule (ICAM), E-selectin, von Willebrand factor | 12 weeks
Fasting lipid profile including measures of total, low density lipoprotein (LDL) and high density lipoprotein (HDL) cholesterol, triglycerides and non-esterified fatty acids | 12 weeks
Indices of insulin resistance derived from fasted measures of glucose, insulin and non-esterified fatty acids (revised QUICKI statistical analysis) | 12 weeks
Haemostatic factors including Plasminogen activator inhibitor-1 (PAI-1) | 12 weeks
Inflammatory biomarkers including the acute phase proteins, C-reactive protein (CRP), tumour necrosis factor alpha (TNFα), Interleukin-6 (IL6) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Commane, PhD, Principal Investigator — Reading University
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Reading, Berkshire, United Kingdom